CLINICAL TRIAL: NCT01353352
Title: Evaluation of the Safety of C-Spine Clearance by Emergency Department Triage Nurses (Phase IV)
Brief Title: Evaluation of the Nursing C-Spine (Phase IV)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ottawa Hospital Research Institute (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Dr Ian Stiell, Principal Investigator, Ottawa Hospital Research Institutute & University of Ottawa
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MOP-86709; 2007542-01H (Other: Ottawa Hospital REB)
Record Dates: First submitted 2010-10-13; First posted 2011-05-13 (Estimated); Last update posted 2011-05-13 (Estimated); Status verified 2011-05

CONDITIONS: Fracture of Cervical Spine; Fracture Dislocation of Cervical Spine
Keywords: Evaluation; C-Spine; Nursing; Clinical Decision Rule

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Cervical spine injury (Other): We enrolled consecutive alert adults who were in stable condition and who presented with potential cervical spine injury after acute blunt trauma, including patients with posterior neck pain and those presenting by ambulance with immobilization of the cervical spine.
  Interventions: Other: Clinical decision rule - clearing the c-spine

INTERVENTIONS:
Other: Clinical decision rule - clearing the c-spine — The goal of phase IV of the Canadian C-Spine Rule project is to evaluate the safety and potential impact of an active strategy to empower ED triage nurses to evaluate and clear the c-spine of very low-risk trauma patients.

SUMMARY:
Neck injuries are a common problem among blunt trauma victims with more than 8,000,000 cases being seen annually in U.S. and Canadian EDs. While the majority of these cases represent soft tissue injuries, 30,000 patients suffer cervical spine fractures or dislocations and approximately 10,000 suffer spinal cord injury. There are no readily available national Canadian data on ED visits such as those provided by the U.S. National Hospital Ambulatory Medical Care Survey. The prevalence of potential neck injury can, however, be reasonably estimated for Canadian EDs. Extrapolation, on a population basis, from reliable U.S. figures suggests that 1.3 million potential neck injury patients are seen annually in Canada. Only 0.9% of these patients are found to have cervical spine fractures or dislocations.

DETAILED DESCRIPTION:
Background: Canadian emergency departments (EDs) annually treat 1.3 million patients who have suffered blunt trauma from falls or motor vehicle collisions and who are at risk for cervical spine injury. Most such cases are alert and stable adults and less than 1% has a c-spine fracture. Most trauma victims transported in ambulances are protected by a backboard, collar, and sandbags and, on arrival at the ED, are sent to high acuity resuscitation rooms, where they remain fully immobilized for hours until physician assessment and radiography are complete. This prolonged immobilization is often unnecessary and adds considerably to patient discomfort and also adds to the burden of our overcrowded Canadian EDs in an era when they are under unprecedented pressures. These patients use valuable ED resuscitation room space.

Nurses usually do not evaluate the c-spine of trauma patients but the investigators believe that they should be able to safely assess alert and stable ambulance patients and "clear" the c-spine of low-risk cases on arrival at the triage station. Patients could then be much more rapidly, comfortably, and efficiently managed in other areas of the ED. An expanded role for nurse decision-making has the potential to improve trauma care efficiency in all Canadian hospitals. Very little research has been done in this area of nurses' clearing patient c-spines.

A clinical decision rule is derived from original research and is defined as a decision making tool that incorporates three or more variables from the history, examination, or simple tests. This Canadian C-Spine Rule (CCR) is comprised of simple clinical variables and was designed to allow clinicians to "clear" the c-spine without radiography and to decrease immobilization times. The investigators also validated the accuracy of the rule when used by physicians. The investigators have now finished a funded study to validate the accuracy and reliability of the CCR when used by ED triage nurses at 6 hospitals. The investigators completed a funded implementation trial at 12 Canadian hospitals to evaluate the impact on patients of the CCR when used by physicians.

Objectives: The goal of phase IV of the Canadian C-Spine Rule project is to evaluate the safety and potential impact of an active strategy to empower ED triage nurses to evaluate and clear the c-spine of very low-risk trauma patients. Specific objectives are to: 1) Determine safety by screening for: a) Missed fractures and b) Serious adverse outcomes; 2) Determine clinical impact by measuring: a) C-spine clearance rates by nurses, b) Length of time until c-spine clearance; 3) Evaluate performance of the Canadian C-Spine Rule for: a) Accuracy, b) Nurse accuracy in interpretation, and c) Nurse comfort and compliance.

Methods: The investigators propose a cohort study which evaluates outcomes during a 12-month period at 5 hospital EDs, including 3 community and 2 teaching hospital sites. Enrolled will be consecutive, alert and stable adult trauma patients presenting to the ED with neck pain or with c-spine immobilization on an ambulance stretcher. Participating will be ED triage nurses who previously underwent a structured educational strategy to learn the CCR and who successfully participated in the 24-month phase IIb validation study at the same sites. These nurses will be empowered by medical directive to "clear" the c-spine of patients according to the CCR, thus allowing them to remove c-spine immobilization and to triage patients to a less acute area of the ED. These outcomes will be assessed: 1) Measures of safety: a) Number of missed fractures, b) Number of serious adverse outcomes; 2) Measures of clinical impact: a) C-spine clearance rates by nurses, b) Length of stay in ED, and c) Patient satisfaction; 3) Performance of the Canadian C-Spine Rule: a) Accuracy, b) Nurse accuracy of interpretation, and c) Nurse comfort. The investigators estimate a sample size of 1,500 patients will be accrued.

Importance: This evaluation study (phase IV) is an essential step in the process of developing a new clinical decision rule / guideline for nurses to clear the c-spine. Once the investigators have established safety and potential impact in phase IV, the investigators can move to the final step (phase V), a multicenter implementation across Canada to study actual impact. The investigators believe that teaching ED triage nurses to clear the c-spine of very low-risk trauma patients has the potential to significantly improve the efficiency and comfort of patient care in our busy Canadian EDs. Ultimately, the investigators expect the results of this study to be used by ED triage nurses throughout Canada.

ELIGIBILITY:
Inclusion Criteria:

The investigators will enroll consecutive alert, stable adults presenting to the study hospital EDs with potential c-spine injury after sustaining acute blunt trauma. These will be patients presenting with neck pain or with c-spine immobilization on an ambulance stretcher. Patient eligibility will be determined based on these criteria at the time of arrival in the ED.

* "Potential c-spine injury after sustaining acute blunt trauma" will include patients with either: i) neck pain with any mechanism of injury (subjective complaint by the patient of any pain in the posterior aspect of the neck), and/or ii) presentation by ambulance with c-spine immobilization after injury (typically backboard and collar).
* "Alert" is defined as a Glasgow Coma Scale103 score of 15 (converses, fully oriented, and follows commands).
* "Stable" refers to normal vital signs as defined by the Revised Trauma Score31 (systolic blood pressure 90 mm Hg or greater and respiratory rate between 10 and 24 breaths per minute).
* "Acute" refers to injury within the past 48 hours.

Exclusion Criteria:

* Patients under the age of 16 years,
* Patients who do not satisfy the definition of "potential c-spine injury" as defined above (for example, patients with neither neck pain nor arriving with ambulance c-spine immobilization will be excluded),
* Patients with Glasgow Coma Scale score less than 15,
* Patients with unstable vital signs (systolic BP < 90; respiratory rate less than 10 or more than 24),
* Patients whose injury occurred more than 48 hours previously,
* Patients with penetrating trauma from stabbing or gunshot wound,
* Patients with acute paralysis (paraplegia, quadriplegia),
* Patients with known vertebral disease (ankylosing spondylitis, rheumatoid arthritis, spinal stenosis, or previous cervical spine surgery),
* Patients who return for reassessment of the same injury, or
* Patients referred from another hospital.

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 3633 (Actual)
Dates: Start 2008-01; Primary Completion 2010-07 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
Determine safety: Number of missed CSI & Number of serious adverse outcomes Determine clinical impact: C-spine clearance rates by nurses & Lengths of time | Dec 2010

SECONDARY OUTCOMES:
Evaluate performance: Accuracy of the rule, Nurse accuracy in overall interpretation of the rule & Nurse comfort with and use of the rule. | Dec 2010
Evaluate performance | December 2010
  Evaluate performance: Accuracy of the rule, Nurse accuracy in overall interpretation of the rule & Nurse comfort with and use of the rule.

CONTACTS AND LOCATIONS:
Overall Officials: Ian G Stiell, MD, Principal Investigator — Ottawa Hospital Research Institute
Locations (1):
- The Ottawa Hospital, Ottawa, Ontario, Canada